CLINICAL TRIAL: NCT05956769
Title: Comparison of TEG-guided and Preemptive Tranexamic Acid Administration Strategies in Total Hip Replacement Surgery
Brief Title: Goal-directed vs Preemptive Tranexamic Acid Administration in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HI22C195200-1-2
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Arthritis of Hip
MeSH Terms: interventions — Tranexamic Acid; Thrombelastography; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomized prospective double-blind placebo-controlled multicenter non-inferior
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Empirical 2: TXA administration (Active Comparator): Tranexamic acid administration, regardless of the result of TEG6.
  Interventions: Drug: Tranexamic Acid; Diagnostic Test: thromboelastography
- Goal-directed 1: Placebo administration (Experimental): Normal saline administration, according to the result of TEG6. . Placebo administration, at LY30 < 3% or MA > 54 mm in CRT of TEG6
  Interventions: Diagnostic Test: thromboelastography; Drug: Placebo
- Goal-directed 2: TXA administration (Experimental): Tranexamic acid administration, according to the result of TEG6. Placebo discard, at LY30> 3% or MA<54 mm in CRT of TEG6
  Interventions: Drug: Tranexamic Acid; Diagnostic Test: thromboelastography

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid injection 10 mg/kg and infusion 2 mg/kg/hr
  Arms: Empirical 2: TXA administration; Goal-directed 2: TXA administration
Diagnostic Test: thromboelastography — thromboelastography (TEG6)
Drug: Placebo — Normal saline injection
  Other Names: Normal saline
  Arms: Goal-directed 1: Placebo administration

SUMMARY:
The present study is a multi-center randomized prospective placebo-controlled non-inferiority trial. The study's primary objective is to compare the amounts of postoperative bleeding using two different TXA administration strategies: empirical TXA administration vs. viscoelastic test-based Goal-directed vs Preemptive Tranexamic Acid Administration in total hip arthroplasty. The secondary objectives include comparing the incidents of hyper-fibrinolysis, thromboembolic complications, and postoperative seizures. Researchers assumed that goal-directed tranexamic acid (TXA) administration using viscoelastic field tests would not be inferior to the empirical TXA administration strategy in reducing postoperative bleeding and hyper-fibrinolysis. It also would be beneficial in lowering TXA-induced thromboembolic complications and seizures.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria patients undergoing following surgery

- total hip arthroplasty

Exclusion Criteria:

* pregnancy
* refusal of allogenic blood transfusion
* taking thrombin
* history of thromboembolic and familial hypercoagulability disease
* recent history of myocardial infarction or ischemic cerebral infarction (within 90 days)
* hypersensitive to TXA
* histroy of convulsion or epilepsy
* taking hemodialysis
* history of Heparin-induced thrombocytopenia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CRT maximal amplitude | 24 hours
  maximal amplitude of CRT test

SECONDARY OUTCOMES:
CK reaction time | 24 hours
  r-time of CRT test
CK alpha angle | 24 hours
  alpha angle of CRT test
CRT maximal lysis | 24 hours
  maximal lysis of CRT test
CFF maximal amplitude | 24 hours
  maximal amplitude of CFF test
Hemoglobin | 6 hours
  the lowest hemoglobin value before transfusion
packed RBC | 6 hours
  transfused fresh frozen plasma
fresh frozen plasma | 6 hours
  transfused fresh frozen plasma
cryoprecipitate | 6 hours
  transfused cryoprecipitate
platelet | 6 hours
  transfused platelet (apheresis) or platelet concentrate
seizure | 48 hours
  postoperative incidence of seizure
thromboembolism | 48 hours
  preoperative incidence of myocardial infarction, cerebral infarction, pulmonary thrombosis, intestinal infarction
postoperative bleeding | 48 hours
  bleeding from surgical drain
re-operation | 48 hours
  re-operation due to postoperative bleeding
intraoperative bleeding | 4 hours
  amount of intraoperative bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Konkuk University Medical Center, Seoul
  - Soi Lee, Seoul

IPD SHARING:
Plan to Share IPD: Undecided